CLINICAL TRIAL: NCT07282262
Title: An Exploratory Study on the Use of Ivosidenib for the Precise Treatment of Advanced Biliary Tract Malignancies With IDH1 Mutations in the Later Line of Therapy.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBLF001
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — ivosidenib; lenvatinib; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Ivosidenib Monotherapy (Experimental)
  Interventions: Drug: Ivosidenib
- Ivosidenib + Lenvatinib (Experimental)
  Interventions: Drug: Ivosidenib; Drug: Lenvatinib
- Ivosidenib + PD-1/PD-L1 Inhibitor (Experimental)
  Interventions: Drug: Ivosidenib; Biological: PD-1/PD-L1 inhibitor
- Ivosidenib + Lenvatinib + PD-1/PD-L1 Inhibitor (Experimental)
  Interventions: Drug: Ivosidenib; Drug: Lenvatinib; Biological: PD-1/PD-L1 inhibitor

INTERVENTIONS:
Drug: Ivosidenib — Oral, selective, small-molecule inhibitor of the mutant isocitrate dehydrogenase 1 (IDH1) enzyme. Administered at a dose of 500 mg, taken orally once daily. This is the core investigational drug in all study arms.
Drug: Lenvatinib — Oral, multi-targeted tyrosine kinase inhibitor. Administered at a weight-based dose (8 mg for body weight <60 kg or 12 mg for body weight ≥60 kg), taken orally once daily. Used in combination arms.
  Arms: Ivosidenib + Lenvatinib; Ivosidenib + Lenvatinib + PD-1/PD-L1 Inhibitor
Biological: PD-1/PD-L1 inhibitor — Intravenous immune checkpoint inhibitor. Specific agent (e.g., Pembrolizumab, Durvalumab, Toripalimab, or Tislelizumab) may be chosen based on local availability and patient access. Administered at standard doses (e.g., 200 mg, 1500 mg, or 240 mg) via IV infusion every three weeks. Used in combination arms.
  Arms: Ivosidenib + Lenvatinib + PD-1/PD-L1 Inhibitor; Ivosidenib + PD-1/PD-L1 Inhibitor

SUMMARY:
This is a multicenter, non-randomized, umbrella, open-label phase II clinical study, aiming to observe and evaluate, as well as explore the efficacy and safety of precision targeted therapy based on NGS technology for IDH1-mutated patients, specifically the combination of ivosidenib with multi-target tyrosine kinase inhibitors represented by lenvatinib or PD-1/PD-L1 in advanced biliary tract cancer patients who have failed systemic chemotherapy.

ELIGIBILITY:
Inclusion Criteria

* Voluntary Participation: Signed informed consent.
* Genetic Mutation: Presence of an IDH1 mutation confirmed by genetic testing.
* Disease Status：
* Newly diagnosed, untreated advanced/metastatic disease; OR
* Recurrence >6 months after curative-intent surgery (with or without adjuvant therapy).
* Measurable Disease: At least one measurable lesion per RECIST 1.1.
* Performance Status: ECOG performance status of 0 or 1.
* Life Expectancy： ≥3 months.
* Organ Function: Adequate hematological, hepatic, and renal function.
* Contraception: Use of highly effective contraception for women of childbearing potential and men.

Exclusion Criteria

* Prior Treatment: Previous treatment with Ivosidenib.
* Cancer Type: Ampulla of Vater cancer.
* Pregnancy： Pregnant or breastfeeding women.
* Allergy: Known hypersensitivity to any component of the study drugs.
* Recent Therapy: Local anti-tumor therapy or major surgery within 4 weeks prior to initiation.
* Medical Conditions:
* Uncontrolled hypertension.
* Significant cardiovascular disease.
* Active or untreated CNS metastases.
* Active autoimmune disease.
* Uncontrolled active infection (e.g., HBV, HCV, HIV).
* Significant bleeding tendency or history.
* Severe non-healing wounds.
* History of organ transplantation.
* Concurrent Participation: Participation in another interventional clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From first dose of study drug until disease progression, death, or start of new anti-cancer therapy, assessed up to approximately 24 months.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | From first dose of study drug until disease progression, death, or start of new anti-cancer therapy, assessed up to approximately 24 months.
Progression-Free Survival (PFS) | From first dose of study drug until disease progression or death from any cause (whichever occurs first), assessed up to approximately 24 months.
Overall Survival (OS) | From enrollment (or first dose) until death from any cause, assessed up to approximately 36 months.
Duration of Response (DOR) | From the date of first documented response (CR or PR) until the date of disease progression or death, assessed up to approximately 24 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Peking Union Medical College Hospital Outpatient Department, Beijing, China

IPD SHARING:
Plan to Share IPD: No